CLINICAL TRIAL: NCT05121441
Title: A Phase 2, Placebo-Controlled, Randomized, Blinded Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of ARD-101 in Adults With Obesity
Brief Title: Study to Evaluate ARD-101 in Adults With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AARD-201
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Obesity; Anti-Obesity Agents; Body Weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: This study includes two arms: one placebo arm and one intervention arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARD-101 (Experimental): Dose 200 mg of ARD-101, twice daily for 28 days
  Interventions: Drug: ARD-101
- Placebo Comparator (Placebo Comparator): Placebo arm matching active arm ARD-101, 200 mg BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARD-101 — Twice daily, oral administration
  Arms: ARD-101
Drug: Placebo — Twice daily, oral administration
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of twice-daily ARD-101 in obese subjects with a body mass index (BMI) of 30-45 kg/m2.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, placebo-controlled study to investigate the effects of ARD-101, a small molecule targeting bitter taste receptors (TAS2Rs), in obese subjects with a body mass index (BMI) of 30-45 kg/m2. This study has a planned enrollment of 30 subjects and will be conducted in a single center in the United States.

The study will consist of a Screening Period (up to 28 days), a Treatment Period (28 days), and a Follow-up Period (End-of-Study Visit within 14 days after receiving the last dose of ARD-101). The screening procedures will be initiated upon completion of the informed consent process. Following completion of screening procedures and confirmation of eligibility, subjects will be enrolled to receive ARD-101 in an outpatient setting and will be instructed to visit the clinical center periodically for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18-75 years of age
* Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures
* BMI of 30-45 kg/m2
* Stable body weight by subject report (± 5%) in the previous 6 months prior to randomization
* No abnormal findings or abnormalities of clinical significance in vital signs, physical examination, clinical laboratory tests (complete blood count (CBC), urinalysis, blood biochemistry, coagulation, pregnancy test (females of child bearing potential), urine drug test, nicotine test, etc.), 12-lead electrocardiogram (ECG) during the Screening Period.
* Serum creatinine, alkaline phosphatase, hepatic enzymes (aspartate aminotransferase, alanine aminotransferase) and total bilirubin (unless the subject has documented Gilbert syndrome) not exceeding 1.5-fold the upper laboratory norm and estimated glomerular filtration rate (eGFR) >30 mL/min
* Standard 12-lead ECG parameters after 10 minutes resting in supine position in the following ranges; 120 ms <PR <220 ms, QRS <120 ms, QTc ≤ 430 ms if male, ≤ 450 ms if female, and normal ECG tracing unless the Investigator considers an ECG abnormality within described limits to be not clinically relevant
* Stable or well controlled blood pressure per Investigator's judgement during the Screening Period. Specifically: Vital signs after 10 minutes sitting in a chair (feet on floor, back supported):

  i. 95 mmHg <systolic blood pressure (SBP) <160 mmHg, ii. 45 mmHg <diastolic blood pressure (DBP) <100 mm Hg, iii. 40 bpm <heart rate (HR) <100 bpm
* Prediabetes- defined as a fasting blood glucose between 100-125 mg/dL OR an HbA1c between 5.7-6.5% at screening
* Type 2 diabetes- Defined as previous diagnosis by a healthcare professional OR a fasting blood glucose > 126 mg/dL OR HbA1c > 6.5% at screening
* Patients with type 2 diabetes treated with metformin may be enrolled. However, patients with type 2 diabetes on any other therapy will be excluded
* Female subjects must have negative serum pregnancy test and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single barrier method (i.e., sponge), or a double-barrier method of birth control (i.e., condom with spermicide) or abstinence must be used/practiced throughout the study and for 90 days following last dose of study medication; for effective form of birth control
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, bilateral tubal ligation, bilateral salpingectomy, or bilateral tubal occlusion) or post-menopausal for at least 12 months (may be confirmed with a screening follicle stimulating hormone (FSH) level in the post-menopausal lab range), do not require contraception during the study
* Males with female partners of childbearing potential must agree to a double-barrier method if they become sexually active during the study and for 90 days following the last dose of the study medication. Male subjects must not donate sperm for 90 days following their participation in the study

Exclusion Criteria:

* History of significant drug hypersensitivity or anaphylaxis
* Prior bariatric or GI surgery (excluding cholecystectomy, hysterectomy or appendectomy)
* Participation in a weight loss program or clinical trial for weight loss within 30 days prior to randomization
* Diabetes treatment (unless metformin as outlined), or chronic oral steroids, or treatment with immune modulators, anti-obesity drugs, chronic opiate therapy, or antipsychotic medications
* Received any experimental drugs or devices or have participated in a clinical study within 30 days prior to randomization
* Currently receiving any drug-based therapy for weight management
* Thyroid-stimulating hormone (TSH) level is outside of normal limit
* The presence of diseases with abnormal clinical manifestations that need to be excluded based on their possible contribution to weight loss or weight gain, including but not limited to nervous, cardiovascular, blood and lymphatic system, immune, renal, hepatic, gastrointestinal, respiratory, metabolic and skeletal diseases
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attack within 6 months prior to Visit 1
* Any malignancy not considered cured (except focal, treated basal cell carcinoma and squamous cell carcinoma of the skin); a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years
* History of major depressive disorder or history of other severe psychiatric disorders (e.g., schizophrenia or bipolar disorder) within the last 2 years.
* Major surgery within 3 months prior to randomization or planned surgery during the study
* Donated ≥200 mL of blood (blood components) or had massive blood loss, received blood transfusion or blood products within 3 months prior to randomization
* Planned sperm/egg donation within 6 months post randomization
* Positive urine drug test for any illicit non-prescription substances
* History of consuming more than 14 units of alcoholic beverages per week or of alcoholism or drug/chemical/substance abuse within past 2 years prior to enrollment (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* Smoking any amount within 3 months prior to randomization
* Excessive consumption of tea, coffee, and/or caffeinated beverages (more than 8 cups, 250 mL for each cup) every day within 3 months prior to enrollment
* Symptomatic viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to randomization
* History of human immunodeficiency virus antibody or active hepatitis
* A history of psychiatric and psychological condition that, in the judgment of the investigator, may interfere with the planned treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications
* Poor venous access or inability to tolerate venipuncture
* Any condition or active drug treatment that the investigator or primary physician believes may not be appropriate for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translational Research Institute, University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referrals at the clinical site between November 2021 and August 2022. A total of 30 subjects were originally planned, but only 20 subjects were enrolled, treated, and analyzed. The first participant was enrolled on November 15, 2021, and the last participant was enrolled in August 2022.
Pre-assignment Details: A total of 20 subjects were enrolled and all 20 (100%) subjects completed the study.
Period: Overall Study
Arm/Group | ARD-101 | Placebo Comparator
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARD-101 | Placebo Comparator | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12) | 49 (9) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kg] | 95.4 (12.4) | 101.6 (23.8) | 97.3 (16.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.1 (3.6) | 35.2 (5.5) | 34.5 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Body Weight (%)
Description: The percent total weight change at the end of treatment from baseline
Time Frame: Run-in Visit (baseline), Day 28
Measure: Mean (Standard Deviation); unit: Percentage of body weight change
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
Percentage of body weight change | -0.33 (0.94) | 0.38 (1.08)

2. Secondary Outcome: Incidence (Number) of Treatment-emergent Adverse Events (TEAE)
Description: The number of treatment-emergent adverse events (TEAE) reported by participants during the treatment period
Time Frame: Days 1-28
Measure: Count of Participants; unit: Participants
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
Participants
  Acid reflux | 1 | 0
  Nausea | 1 | 0
  No TEAE reported | 12 | 6

3. Secondary Outcome: Change in TC
Description: The change in total cholesterol (TC) at the end of treatment from baseline
Time Frame: Days 1 to 28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
mg/dL | -4.4 (17.32) | 5.7 (19.31)

4. Secondary Outcome: Change in TG
Description: The change in triglyceride (TG) at the end of treatment from baseline
Time Frame: Days 1-28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
mg/dL | -0.6 (93.81) | 0.5 (27.60)

5. Secondary Outcome: Change in HDL
Description: The change in high density lipoprotein cholesterol (HDL) at the end of treatment from baseline
Time Frame: Days 1-28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
mg/dL | 0.2 (7.36) | 4.0 (6.10)

6. Secondary Outcome: Change in LDL
Description: The change in low-density lipoprotein cholesterol (LDL) at the end of treatment from baseline
Time Frame: Days 1-28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 13 | 6
mg/dL | -6.8 (16.95) | 1.3 (15.15)

7. Secondary Outcome: Change in Waist Circumference
Description: The change in waist circumference at the end of treatment from baseline
Time Frame: Days 1-28
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
cm | -0.2 (1.7) | -0.8 (3.3)

8. Secondary Outcome: Change in % HbA1C
Description: The change in % of hemoglobin A1c (HbA1c) at the end of treatment from baseline
Time Frame: Screening to Day 28
Measure: Mean (Standard Deviation); unit: Percent of HbA1c
Arm/Group | ARD-101 | Placebo Comparator
Number analyzed (Participants) | 14 | 6
Percent of HbA1c | -0.17 (0.22) | -0.18 (0.24)

ADVERSE EVENTS:
Time Frame: Six weeks (28-day treatment period plus 14-day follow-up post treatment)
Arm/Group | ARD-101 | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 3/14 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARD-101 (N=14) | Placebo Comparator (N=6)
Acid Reflux (Gastrointestinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Foot Injury (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT05121441/Prot_SAP_000.pdf